CLINICAL TRIAL: NCT03426553
Title: Clinical Application of Red Blood Cell Suspension, Obtained From the Pathogen Reduced Whole Blood in Children With Oncological and Hematological Diseases
Brief Title: Clinical Use of Pathogen Reduced Red Blood Cell Suspension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Rb+UV_WB_01_2017
Record Dates: First submitted 2017-10-10; First posted 2018-02-08 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Oncologic Disorders; Hematologic Diseases
Keywords: Patogen inactivation; Pathogen reduction; clinical use; riboflavin+UV; RBC transfusion; whole blood
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Riboflavin+UV RBC (Experimental): 35 patients who met all inclusion and exclusion criteria received transfusion with RBC suspension from whole blood, treated with riboflavin and ultraviolet pathogen reduction technology
  Interventions: Biological: Riboflavin+UV RBC
- irradiated RBC (Active Comparator): 35 patients who met all inclusion and exclusion criteria received transfusion with irradiated RBC suspension
  Interventions: Biological: irradiated RBC

INTERVENTIONS:
Biological: Riboflavin+UV RBC — 35 patients who met all inclusion and exclusion criteria received transfusion with RBC suspension from whole blood, treated with riboflavin and ultraviolet pathogen reduction technology
  Arms: Riboflavin+UV RBC
Biological: irradiated RBC — 35 patients who met all inclusion and exclusion criteria received transfusion with irradiated RBC suspension
  Arms: irradiated RBC

SUMMARY:
The aim of the study is to evaluate the effectiveness and safety of the application of pathogen inactivated RBC suspension in children with oncological and hematological diseases.

DETAILED DESCRIPTION:
Assumed scope of study:

The study will include 70 patients: 35 patients to the test group, who will get transfusions with pathogen-inactivated red blood cell suspension; 35 patients to the control group, who will get transfusions with irradiated red blood cell suspension.

Methods:

* Selection of patients suitable to participate in the study.
* A few days before the assumed transfusion date, select/prepare a red blood cell suspension corresponding to ABO and Rh systems, with no more than 14 days of storage. Conduct direct antiglobuline test (DAT), indirect antiglobuline test (IAT) and test for individual compatibility with the patient's serum.
* Before performing transfusion (on the day of transfusion), determine the initial indices of the patient (Hb, Hct, Haptoglobin). Determine the red blood cell suspension indices (Hb, Hct, extracellular potassium, free hemoglobin, hemolysis percentage).
* Perform transfusion. Evaluate the presence and severity of post-transfusion reactions and complications.
* Measure the patient's Hb, Hct, potassium and haptoglobin levels the next day after the transfusion.
* Perform DAT 3 to 5 five days after the transfusion.
* Perform IAT 2 to 3 weeks after the transfusion.
* Evaluate the need for transfusions over the follow-up period (30 days).

ELIGIBILITY:
Inclusion Criteria:

Patients who need supportive transfusion therapy with RBC suspension

Exclusion Criteria:

* Active bleeding
* Sepsis/severe infection (any infectious disease requiring pressor agents, infusion and respiratory support)
* Positive DAT and / or IAT before transfusion
* Double populations for ABO and RH blood group antigens
* Severe hepatomegaly/splenomegaly
* Patients receiving chemotherapy (at the time of need for transfusion)
* Patients receiving antithymocyte immunoglobulin and also within 7 days after its completion
* Patients requiring transfusion of only irradiated blood components

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-09-17 (Actual); Study Completion 2018-12-17 (Actual)

PRIMARY OUTCOMES:
post-transfusion reactions | 24 hours after transfusion
  evaluate the presence and severity of post-transfusion reactions and complications.
augmentation of hemoglobin | 24 hours after transfusion
  Measure the patient's hemoglobin concentration (g/dL) the next day after the transfusion
augmentation of hematocrit | 24 hours after transfusion
  Measure the patient's hematocrit (%) the next day after the transfusion
immune responses | 3-5 days after transfusion
  Perform direct antiglobuline test
sensitization | 2-3 weeks after transfusion
  perform indirect antiglobuline test
intertransfusion interval | 1 months
  Evaluate the need for transfusions over the follow-up period (30 days)

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Trakhtman, PhD, Study Director — Federal Research Center for pediatric hematology, oncology and immunology
Locations (1):
- Federal Research Center for pediatric hematology, oncology and immunology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No